CLINICAL TRIAL: NCT06812897
Title: Assessing the Feasibility of a Patient-Driven Chiropractic Patient Portal (SallieTM Life U) for Research Purposes
Brief Title: Sallie Life U Feasibility Study
Acronym: SLU
Status: Active, not recruiting | Type: Observational
Sponsor: Life University (Other)
Collaborators: Power of Patients (Unknown)
Responsible Party: Sponsor
Other Study IDs: I-0031
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy: Healthy subjects
  Interventions: Other: Sallie (TM) Life U

INTERVENTIONS:
Other: Sallie (TM) Life U — Testing of Sallie (TM) Life U platform

SUMMARY:
This feasibility trial explored the usability of the patient-driven chiropractic patient portal, Sallie™ Life U. The study aimed to recruit 30 participants to track their daily symptoms, triggers, and habits over 30 days while completing three questionnaires about their experience with the portal. The first questionnaire was administered after participants created their accounts, the second at the midpoint of tracking (day 15), and the third upon completing the tracking period (day 30). All participation in the study was conducted remotely using the participants' personal devices.

ELIGIBILITY:
Inclusion Criteria:

* Have daily access to technology (smartphone, tablet, or computer)
* Currently receiving chiropractic care (for the purposes of this feasibility study, this requires at least one chiropractic adjustment each month)

Exclusion Criteria:

- Given software restrictions, participants must also be able to read and write in English and not be visually impaired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No specific population
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment | 30 days
  Average # of participants to create a SallieTM Life U account per month
Participant Adherence - Weekly | 30 days
  % of participants with daily data input throughout the week
Participant Adherence - Monthly | 30 days
  % of participants with total number of daily data input throughout the month.
Participant Retention | 30 days
  % of participants completing all questionnaires

SECONDARY OUTCOMES:
Personalized Tracking Metrics (PTMs) | 30 days
  Self-generated habits or personal goals that participants create and track in their portals

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, PhD, Study Director — Dr. Sid E Williams Center for Chiropractic Research
Locations (1):
- Dr. Sid E Williams Center for Chiropractic Research, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No